CLINICAL TRIAL: NCT01968941
Title: A Randomized Trial of Medically-Inoperable Stage 1 Non-small Cell Lung Cancer Patients Comparing Stereotactic Body Radiotherapy Versus Conventional Radiotherapy
Brief Title: Stereotactic Body Radiotherapy Versus Conventional Radiotherapy in Medically-Inoperable Non-Small Lung Cancer Patients
Acronym: LUSTRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2013-LUSTRE
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: stereotactic body radiotherapy; conventional radiotherapy; inoperable patients; local control; cancer recurrence; toxicity; survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiotherapy (Experimental): Stereotactic Body Radiotherapy (SBRT)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Conventional Radiotherapy (Active Comparator): Conventional Radiotherapy (CRT)
  Interventions: Radiation: Conventional Radiotherapy (CRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT)
  Arms: Stereotactic Body Radiotherapy
Radiation: Conventional Radiotherapy (CRT)
  Arms: Conventional Radiotherapy

SUMMARY:
A multi-centre randomized controlled open-label trial in medically inoperable patients with biopsy-proven early stage non-small cell lung cancer (NSCLC). Eligible and consenting patients will be randomly allocated to receive stereotactic body radiotherapy (SBRT) or conventional radiotherapy (CRT) in a 2:1 ratio. Radiotherapy will be administered as soon as possible following randomization and subjects will be followed for 5 years post-randomization for cancer recurrence, toxicity and survival. The primary outcome is local control (LC). The trial will be conducted at 16-20 clinical centres throughout Canada.

ELIGIBILITY:
Inclusion Criteria:

1. T1/T2a N0 M0 NSCLC, either by: (a) histological confirmation (squamous cell, adenocarcinoma, large cell carcinoma, or not specified) and CT thorax and/or PET-CT evidence, or (b) a suspicious growing nodule on serial CT imaging, with malignant PET Fluorodeoxyglucose (FDG) avidity, for which a biopsy would be extremely risky.
2. Deemed medically inoperable (as reviewed by a thoracic surgeon and defined as surgically resectable but, because of underlying physiological medical problems [e.g. chronic obstructive pulmonary disease (COPD), heart disease], surgery is contraindicated) or Radiotherapy is preferred by the patient due to high operable risk.

Exclusion Criteria:

1. Less than 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher.
3. Prior invasive malignancy within the past 3 years (excluding non-melanomatous skin cancer).
4. History of ataxia telangiectasia.
5. Previous radiotherapy (RT) in the vicinity of the tumour, such that significant overlap could occur.
6. Previous pneumonectomy with Stage I lung cancer in the remaining lung.
7. Diagnosis of idiopathic pulmonary fibrosis and/or interstitial lung disease.
8. Planned for other anticancer therapy (chemotherapy, biological targeted therapy).
9. Female, who is currently pregnant or lactating.
10. Geographic inaccessibility for follow-up.
11. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2014-05-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Local Control | 5 years
  Local control is the absence of local recurrence during the study period. This is the time from randomization to primary tumour failure or marginal failure.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall Survival is defined as the time from randomization to death from any cause. Alive subjects will be censored on the date of last follow-up.
Disease-Free Survival | 5 years
  Disease-Free Survival is defined as the time from randomization to the earliest recurrence of disease or to death attributed to lung cancer.
Event-Free Survival | 5 years
  Event-Free Survival is defined as the time from randomization to the earliest documented recurrent disease or death from any cause.
Lung Cancer-Specific Survival | 5 years
  Lung Cancer-Specific Survival is defined as the time from randomization to death attributable to lung cancer
Radiation Treatment-Related Death | 1 to 12 months
  Radiation Treatment-Related Death is defined as death occurring between 1 to 12 months following treatment, and caused directly by radiation toxicity attributed to either catastrophic hemorrhage or to severe radiation pneumonitis leading to death
Toxicity | 5 years
  Acute Toxicity will be assessed at 3 months post-randomization and includes fatigue, dyspnea and esophagitis. Late toxicity will be assessed beyond 3 months and up to 5 years and includes radiation pneumonitis, chest wall pain and rib fracture.
Quality of Life | 2 years
  Impact on quality of life will be assessed with the European Organization for Research in Treatment of Cancer and the Lung Cancer-specific Module 13 questionnaires.
Cost-Utility | 3 years
  Cost-Utility will be assessed using the European Quality of Life questionnaire in conjunction with the overall survival results

CONTACTS AND LOCATIONS:
Overall Officials: Anand Swaminath, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Tim Whelan, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (16):
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Horizon Health Network, Saint John, New Brunswick
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at the Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Niagara Health System-Walker Family Cancer Centre, St. Catharines, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Charles LeMoyne Hospital, Greenfield Park, Quebec
  - CHUM Hospital Notre Dame, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Montreal General Hospital McGill, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Rosenberg SA, Mak R, Kotecha R, Loo BW Jr, Senan S. The Nordic-HILUS Trial: Ultracentral Lung Stereotactic Ablative Radiotherapy and a Narrow Therapeutic Window. J Thorac Oncol. 2021 Oct;16(10):e79-e80. doi: 10.1016/j.jtho.2021.06.030. No abstract available. PMID 34561039